CLINICAL TRIAL: NCT06325397
Title: Less Discomfort and Less Pharmacology. Cataract Surgery at Physiologic Intraocular Pressure (IOP)
Status: Completed | Type: Observational
Sponsor: Matthew Rauen (Other)
Responsible Party: Sponsor-Investigator, Matthew Rauen, MD, Wolfe Eye Clinic
Organization: Wolfe Eye Clinic (Other)
Other Study IDs: IIT #88313865
Record Dates: First submitted 2024-01-04; First posted 2024-03-22 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Nuclear Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- High Intraocular Pressure (IOP): Eyes in this arm will maintain an Intraocular Pressure (IOP) of 65 millimeters of mercury (mmHg) throughout the cataract surgery.
  Interventions: Other: High Intraocular Pressure (IOP)
- Low Intraocular Pressure (IOP): Eyes in this arm will maintain an Intraocular Pressure (IOP) of 24 millimeters of mercury (mmHg) throughout the cataract surgery.
  Interventions: Other: Low Intraocular Pressure (IOP)

INTERVENTIONS:
Other: High Intraocular Pressure (IOP) — Prospective, single-surgeon, randomized, paired-eye study; patients undergoing sequential, uncomplicated bilateral phacoemulsification using Active Sentry handpiece® with Intraocular Pressure (IOP) ≤ 24 millimeters of mercury (mmHg) (low IOP) in one eye and with IOP ≥ 65 millimeters of mercury (mmHg) (high IOP) in the other eye.
  Groups: High Intraocular Pressure (IOP)
Other: Low Intraocular Pressure (IOP) — Low Intraocular Pressure (IOP) Prospective, single-surgeon, randomized, paired-eye study; patients undergoing sequential, uncomplicated bilateral phacoemulsification using Active Sentry handpiece® with intraocular IOP ≤ 24 millimeters of mercury (mmHg) (low IOP) in one eye and with IOP ≥ 65 millimeters of mercury (mmHg) (high IOP) in the other eye
  Groups: Low Intraocular Pressure (IOP)

SUMMARY:
To investigate the impact of high vs low Intraocular Pressure (IOP) on the intraoperative experience for the patient and surgeon. Operating at a more physiologic IOP using Active Sentry hand piece during cataract surgery will result in significantly less discomfort/pain as assessed by the decreased need for rescue medication

DETAILED DESCRIPTION:
Objectives:

To investigate the impact of Intraocular Pressure (IOP) high vs low on the intraoperative experience for the patient and surgeon

Design:

Prospective, single-surgeon, subject's first eyes undergoing phacoemulsification will be randomized to high (Intraocular Pressure (IOP) 65 millimeters of mercury (mmHg)) or low (IOP 25mmHg) IOP, contralateral eye will receive other treatment

Hypothesis:

Operating at a more physiologic IOP using Active Sentry hand piece during cataract surgery will result in significantly less discomfort/pain as assessed by the decreased need for rescue medication

ELIGIBILITY:
Inclusion Criteria:

* Visually significant cataract 2-3+ undergoing uncomplicated cataract surgery
* Unremarkable ocular health but inclusive of early Age related macular degeneration (AMD).

Exclusion Criteria:

* History of ocular surgery including corneal refractive surgery
* Compromised zonular integrity or stability
* Uncontrolled diabetes and diabetic retinopathy
* Small pupils
* History of systemic inflammatory disease/uveitis
* History of psychiatric illness, chronic pain/narcotics, benzodiazepine usage
* Abnormal liver or renal function

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 75 cataract surgery patients from ophthalmology clinic
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Medication Rescue | Intraoperative
  Percentage (%) of pts in each group requiring treatment for breakthrough discomfort/pain

SECONDARY OUTCOMES:
Physiologic Responses associated with pain/inflammation: | Intraoperative
  Blood pressure- measured systolic pressure over the diastolic pressure
Physiologic Responses associated with pain/inflammation: | Intraoperative
  Pulse rate- measured in beats per minute (bpm)
Surgeon Experience: Assessment on patient cooperation | Intraoperative
  Surgeon assessment on patient cooperation: poor, good, excellent
  1. Poor cooperation: could not follow instructions, lid squeezing, patient had frequent eye & head movements
  2. Good cooperation: able to follow directions 50% of the time, some lid squeezing and patient movement
  3. Excellent cooperation: able to follow directions >80% of the time with limited lid squeezing and patient movement
Surgeon Experience: Surgeon intraoperative experience | Intraoperative
  Surgeon assessment on overall experience: poor, good, excellent
  1. Poor: fluctuating chamber (reverse pupillary block or surge) and reduced efficiency (nucleus & cortex removal)
  2. Good: >75% chamber stability and adequate efficiency
  3. Excellent: Minimal to no fluctuating chamber and excellent efficiency
Cost- analysis | Intraoperative
  Cost-analysis on intraoperative pharmacological agents utilized between high vs low Intraocular Pressure (IOP)

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfe Eye Clinic, West Des Moines, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gills JP, Cherchio M, Raanan MG. Unpreserved lidocaine to control discomfort during cataract surgery using topical anesthesia. J Cataract Refract Surg. 1997 May;23(4):545-50. doi: 10.1016/s0886-3350(97)80211-8. PMID 9209989
- [Background] Crandall AS, Zabriskie NA, Patel BC, Burns TA, Mamalis N, Malmquist-Carter LA, Yee R. A comparison of patient comfort during cataract surgery with topical anesthesia versus topical anesthesia and intracameral lidocaine. Ophthalmology. 1999 Jan;106(1):60-6. doi: 10.1016/S0161-6420(99)90007-6. PMID 9917782
- [Background] Reddy AJ, Dang A, Dao AA, Arakji G, Cherian J, Brahmbhatt H. A Substantive Narrative Review on the Usage of Lidocaine in Cataract Surgery. Cureus. 2021 Oct 30;13(10):e19138. doi: 10.7759/cureus.19138. eCollection 2021 Oct. PMID 34737914